CLINICAL TRIAL: NCT02414360
Title: Using a Systematic Review in Clinical Decision Making: a Pilot Parallel, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Laure Perrier, PhD Candidate, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 487776
Record Dates: First submitted 2015-04-03; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Evidence-Based Medicine
Keywords: Review Literature as Topic
MeSH Terms: interventions — TAL1 protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shortened Format (Experimental): Shortened format of a systematic review
  Interventions: Other: Shortened Format
- Control (Active Comparator): Full length systematic review
  Interventions: Other: Full Length

INTERVENTIONS:
Other: Shortened Format — Shortened format of a systematic review
  Arms: Shortened Format
Other: Full Length — Full length systematic review
  Arms: Control

SUMMARY:
The purpose of this pilot study is to determine the feasibility of running a full-scale trial that compares two formats of a shortened systematic review to a full-length systematic review to be used in clinical decision-making.

DETAILED DESCRIPTION:
Two shortened systematic review formats were developed to enhance their use in clinical decision making. An online randomized controlled trial is planned to make comparisons of the shortened formats to a full-length systematic review. To prepare for the full-scale trial, a pilot study will be conducted to test methods and procedures in order to refine the processes.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who were in practice full- or part-time at study enrollment were recruited for participation
* Participants had to have access to the Internet as the study was conducted online.

Exclusion Criteria:

* The systematic reviews in all formats were only available in English, thus any participants who were not able to read and understand English were not eligible to participate.
* Anyone who had taken part in any phase of the development of the shortened versions of the systematic reviews (cased-based or evidence-expertise formats) were not eligible for recruitment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessment of participant's answers measured using a kappa statistic | 6 months
  Feasibility of assessing participants' answers
Rate of recruitment | 6 months
  Feasibility of recruiting participants in a timely manner

REFERENCES:
- [Background] Perrier L, Persaud N, Ko A, Kastner M, Grimshaw J, McKibbon KA, Straus SE. Development of two shortened systematic review formats for clinicians. Implement Sci. 2013 Jun 14;8:68. doi: 10.1186/1748-5908-8-68. PMID 23767771
- [Background] Perrier L, Kealey MR, Straus SE. An iterative evaluation of two shortened systematic review formats for clinicians: a focus group study. J Am Med Inform Assoc. 2014 Oct;21(e2):e341-6. doi: 10.1136/amiajnl-2014-002660. Epub 2014 May 1. PMID 24786378
- [Background] Perrier L, Kealey MR, Straus SE. A usability study of two formats of a shortened systematic review for clinicians. BMJ Open. 2014 Dec 23;4(12):e005919. doi: 10.1136/bmjopen-2014-005919. PMID 25537782
- [Derived] Perrier L, Persaud N, Thorpe KE, Straus SE. Using a systematic review in clinical decision making: a pilot parallel, randomized controlled trial. Implement Sci. 2015 Aug 15;10:118. doi: 10.1186/s13012-015-0303-4. PMID 26276278